CLINICAL TRIAL: NCT04965129
Title: Effect of Supplementation of Poly-unsaturated n-3 Fatty Acids and High-protein Diet on Epigenetic Modulation of Muscle Mass, Dose-limiting Toxicity and Intestinal Microbiota in Patients With Lung Cancer Submitted to Treatment With Immunotherapy, Chemotherapy and Tyrosine Kinase Inhibitors.
Brief Title: Supplementation of n-3 PUFA in the Modulation of Lean Mass in Patients With Lung Cancer Receiving a High-protein Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Institutos Madrileño de Estudios Avanzados IMDEA (Unknown); Oncoclínicas (Industry)
Responsible Party: Principal Investigator, Wilza Arantes Ferreira Peres, Associate professor, Institute of Nutrition, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40240420.2.0000.5533
Record Dates: First submitted 2021-05-20; First posted 2021-07-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: fish oils; body composition; microbiota; epigenetics; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: Placebo (Placebo Comparator): Placebo Comparator: Placebo All subjects will be given placebo identically matched with regard to shape, color and taste. They will be given four tablet/day for four mounths.
  Interventions: Drug: Placebo
- Experimental: Fish oil (Experimental): All subjects will be given fish oil with a dose of 2.100 mg of EPA and 924 mg of DHA, in four tablet twice daily for four mounths.
  Interventions: Drug: Fish oil

INTERVENTIONS:
Drug: Placebo — Drug: Placebo olive oil pill manufactured to mimic fish oil. Other Names: • Placebo
  Arms: Placebo Comparator: Placebo
Drug: Fish oil — All subjects will be given fish oil with a dose of of 2.100 mg of EPA and 924 mg of DHA, in four tablet twice daily for four mounths.
  Other Names: Vital Fish
  Arms: Experimental: Fish oil

SUMMARY:
This study is conducted to test the hypothesis that patients with lung cancer undergoing treatment with immunotherapy, chemotherapy and tyrosine Kinase Inhibitors receiving a high protein diet and supplemented with fish oil will improve muscle mass, therapeutic response and modulate the intestinal microbiota within a 4 month period.

DETAILED DESCRIPTION:
Lung cancer (PC) is the most prevalent tumor. The loss of muscle mass, myosteatosis and changes in body composition have been associated with inflammation in cancer and PUFA n-3 have been shown to be an important modulator of the inflammatory response and epigenetic mechanisms. Additionally, the intestinal microbiome has received prominence with the use of immunotherapy, as it is demonstrating that resistance to this therapy can be attributed to the abnormal composition of the intestinal microbiome. Aims: The purpose of this study is to assess the effects of fish oil supplementation in the modulation of lean mass and intestinal microbiome in patients with lung cancer undergoing treatment with immunotherapy, chemotherapy and Tyrosine Kinase Inhibitors receiving a high-protein diet. Methods: Fifty patients will be randomly allocated either to treatment with fish oil or to placebo for 4 months. The following assessments will be made: lean mass, myosteatosis, sarcopenia, adipose compartment, inflammation, micro RNA, food consumption, membrane phospholipid composition, composition of the intestinal microbiota, toxicity, response to antineoplastic treatment and survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small cell lung cancer, both sexes, ECOG performance status (0-2) eligible for treatment with immunotherapy, chemotherapy and tyrosine Kinase Inhibitors.

Exclusion Criteria:

* supplementation of PUFA n-3 in the last 6 months; weight loss> 10% in 6 months, chronic liver disease, previous chronic kidney disease, anorexia, decompensated diabetes mellitus and dementia.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass | 16 weeks
  CT-derived changes in muscle mass ocurring from baseline to week 16

SECONDARY OUTCOMES:
Red blood cell omega-3 fatty acid concentrations (eicosapentaenoic [EPA] and docosahexaenoic acid [DHA] | 16 weeks
  Assessed by gas chromatography (GC)
Muscle strenght | 16 weeks
  Hand grip strength test
Change in fecal microbiome composition | 16 weeks
  alpha- and beta-diversity of 16S bacterial rDNA
Change in levels of miRNA 133 | 16 weeks
  Measure the plasma levels of miRNA 133 from baseline to week 16 by real-time PCR
Change/maintenance in overall skeletal muscle density. | 16 weeks
  To assess the change/maintenance in muscle density from baseline to week 16 using computed tomography (CT).

CONTACTS AND LOCATIONS:
Overall Officials: Wilza AF Peres, PhD, Principal Investigator — Post-graduation in Nutrition, Institute of Nutrition
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No